CLINICAL TRIAL: NCT06816264
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of Oral HRS-5346 in Adult Patients at High Risk of Cardiovascular Events With Elevated Lipoprotein(a)
Brief Title: A Study of HRS-5346 in Adult Participants With Elevated Lipoprotein(a) at High Risk for Cardiovascular Events
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-5346-201
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Treatment of Lipoprotein Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HRS-5346 Dose 1 (Experimental)
  Interventions: Drug: HRS-5346
- HRS-5346 Dose 2 (Experimental)
  Interventions: Drug: HRS-5346
- HRS-5346 Dose 3 (Experimental)
  Interventions: Drug: HRS-5346
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HRS-5346 — HRS-5346
  Arms: HRS-5346 Dose 1; HRS-5346 Dose 2; HRS-5346 Dose 3
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of HRS-5346 in adult participants with elevated Lp(a) at high risk for cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

1. Understanding the specific procedures of the trial, voluntarily participating in this trial, and providing written informed consent;
2. Being at least 18 years of age on the day of signing the informed consent form;
3. Body Mass Index (BMI) within the range of 18.5 to 40 kg/m² (inclusive of boundary values);
4. Participants must be at high risk of cardiovascular events, defined as individuals diagnosed with Atherosclerotic Cardiovascular Disease (ASCVD) and those at high risk for ASCVD.
5. Participants (including their partners) are willing to voluntarily use highly effective contraceptive measures from the time of signing the informed consent form until 6 months after the last administration of the study drug; female participants must have a negative blood pregnancy test and must not be breastfeeding;
6. Willing and able to comply with all the provisions of the protocol, including demonstrating the ability to adhere to study procedures prior to random assignment.

Exclusion Criteria:

- Medical History and Concomitant Medications

1. Occurrence of any of the following events within 3 months prior to screening, or between screening and randomization, or any other event deemed by the investigator to indicate clinical instability: major cardiac or non-cardiac surgery, coronary, carotid, or peripheral artery revascularization, stroke or transient ischemic attack, myocardial infarction or unstable angina, acute limb ischemia;
2. Planned or anticipated cardiac, cerebrovascular, or peripheral artery surgery or coronary revascularization or other major surgery after randomization;
3. History of hemorrhagic stroke or other significant bleeding events;
4. History of malignancy in any organ system (except well-treated basal cell carcinoma of the skin);
5. History of diseases that significantly affect lipid levels, such as nephrotic syndrome, severe liver disease, Cushing's syndrome, etc.;
6. Uncontrolled type 1 or type 2 diabetes within 6 months prior to screening (including diabetic ketoacidosis or hyperosmolar hyperglycemic state or HbA1c > 8.5% at screening);
7. History of acute kidney injury within 12 months prior to screening;
8. Uncontrolled hyperthyroidism or hypothyroidism;
9. Active infection requiring systemic antiviral or antibiotic therapy prior to randomization;
10. New York Heart Association (NYHA) class III-IV heart function or most recent left ventricular ejection fraction (LVEF) < 30% at screening or prior to randomization;
11. Use of weight-loss medications or surgery leading to weight instability within 2 months prior to screening;
12. Long-term continuous or repeated use of systemic corticosteroids within 3 months prior to screening (excluding local use, such as intra-articular, nasal, inhaled, topical, etc.; long-term continuous means ≥7 days; repeated means cumulative use ≥3 times);
13. Lipoprotein apheresis treatment within 3 months prior to screening, or planned to undergo this treatment during the study;
14. Use of PCSK9 inhibitors within 12 months prior to screening;
15. Allergy to the active ingredient of HRS-5346 or any excipient.

    Laboratory and Other Tests
16. Uncontrolled hypertension at screening (sitting systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg);
17. Severe renal insufficiency, defined as eGFR < 30 ml/min/1.73 m² (calculated using the CKD-EPI formula) at screening, or undergoing dialysis;
18. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or γ-glutamyl transferase (GGT) more than 3 times the upper limit of normal (ULN), or total bilirubin more than 2 times the ULN;
19. Positive test results for any of the following: human immunodeficiency virus antibody (HIV-Ab), hepatitis C virus antibody (HCV-Ab), Treponema pallidum antibody; positive hepatitis B virus surface antigen (HBsAg) with HBV-DNA ≥1000 copies/ml (or ≥200 IU/ml, if the lower limit of detection is higher than 1000 copies/ml or 200 IU/ml, then HBV-DNA ≥ the lower limit of detection);
20. Creatine kinase (CK) more than 3 times the ULN;
21. Thyroid-stimulating hormone (TSH) below the lower limit of normal (LLN) or more than 1.5 times the ULN;

    Other Conditions
22. History of drug or alcohol abuse or dependence within the past 1 year;
23. Pregnant or breastfeeding women;
24. Participants in any drug or medical device clinical trial within 3 months prior to screening (defined by the participant receiving the trial drug/device treatment), or within 5 half-lives of the trial drug prior to screening, whichever is longer;
25. Participants deemed by the investigator to have poor compliance or any factors that make them unsuitable for this trial, including but not limited to participation posing unacceptable risk to the participant or potentially interfering with study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2025-02-18 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Percent Change from Baseline in Lipoprotein (a) Lp(a) | Baseline to Week 12

SECONDARY OUTCOMES:
The percentage of all reported adverse events, serious adverse events and treatment-related adverse events, serious adverse events. | From Day 1 to Week 16
Percentage of Participants Achieving Lp(a) <125 Nanomole/Liter (nmol/L) | Week 12
Percentage of Participants Achieving Lp(a) <75 Nanomole/Liter (nmol/L) | Week 12
The plasma concentration of HRS-5346. | From Day 1 to Week 16

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided